CLINICAL TRIAL: NCT04258787
Title: Evaluating Corneal Edema in Fuchs' Endothelial Dystrophy Using Optical Coherence Tomography
Brief Title: OCT in Fuchs' Dystrophy
Status: Recruiting | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, David Huang, Principal Investigator, Oregon Health and Science University
Other Study IDs: OHSU IRB#00020108; R01EY029023-01 (NIH)
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Fuchs Dystrophy; Pseudophakic Bullous Keratopathy
Keywords: Fuchs; Pseudophakic Bullous Keratopathy; Optical Coherence Tomography (OCT); PBK
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group A: No Surgery Group: This group consists of adults ages 18 or older who have been diagnosed with Fuchs' dystrophy or pseudophakic bullous keratopathy but do not require surgery per standard-of-care guidelines.
- Group B: Surgery Group: This group consists of adults ages 18 or older who have been diagnosed with Fuchs' dystrophy or pseudophakic bullous keratopathy, who require Descemet's Stripping Endothelial Keratoplasty (DSAEK), Descemet's Membrane Endothelial Keratoplasty (DMEK), or Descemet's Stripping Only (DSO) surgery. All treatment decisions will be made by the attending physician based on standard-of-care guidelines. (The study does not designate a treatment modality or pay for the treatment.)

SUMMARY:
This is an observational study using optical coherence tomography (OCT) technology to quantify corneal edema in Fuchs' endothelial dystrophy and predict refractive shift from resolving corneal edema after surgical treatments.

ELIGIBILITY:
Inclusion Criteria:

* Damaged or diseased corneal endothelium from Fuchs' or PBK
* Willingness to commit to required study visits

Exclusion Criteria:

* Prior Endothelial Keratoplasty (EK) or any other surgery except uncomplicated cataract surgery
* Presence of a condition that increases the probability for treatment failure (e.g., heavily vascularized cornea, uncontrolled uveitis)
* Other primary endothelial dysfunction conditions (e.g., posterior polymorphous corneal dystrophy and congenital hereditary corneal dystrophy, iridocorneal endothelial syndrome)
* Central sub-epithelial or stromal scarring that could impact post-operative clarity assessment
* Peripheral anterior synechiae in the angle greater than 3 clock hours
* Hypotony
* Uncontrolled glaucoma
* Visually significant optic nerve or macular pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults age 18 or older with Fuchs' or PBK
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-06-26 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Corneal Epithelial Edema/Haze | up to 2 years
  OCT will be used to measure corneal epithelial edema/haze (in microns) in participants with Fuchs' or PBK
Corneal Stromal Edema/Haze | up to 2 years
  OCT will be used to measure corneal stromal edema/haze (in microns) in participants with Fuchs' or PBK

CONTACTS AND LOCATIONS:
Overall Officials: Winston Chamberlain, MD, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No